CLINICAL TRIAL: NCT03847272
Title: A Multicenter Phase 2 Single-arm Proof-of-concept Trial to Assess the Efficacy and Safety of Ustekinumab in Association With Prednisone for the Treatment of Non-infectious Severe Uveitis (NISU)
Acronym: USTEKINISU
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The long inclusion period meant that the question could not be answered within an appropriate timeframe.
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIELEFELD Janssen-PHRC N 2017
Record Dates: First submitted 2019-02-15; First posted 2019-02-20 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Patients With Newly Diagnosed Active NISU
MeSH Terms: interventions — Prednisone; Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental)
  Interventions: Drug: prednisone and ustekinumab treatment; Other: Ophthalmologic examination; Other: Questionnaires; Biological: Blood samples

INTERVENTIONS:
Drug: prednisone and ustekinumab treatment — Treatment with prednisone and ustekinumab (90 mg subcutaneously at inclusion (W0), W4 and W16)
Other: Ophthalmologic examination — Best corrected visual acuity (BCVA) testing, Slit Lamp Exam, tonometry, dilated indirect ophthalmoscopy, optical coherence tomography (OCT), Fluorescein angiography and Indocyanin green angiography
Other: Questionnaires — VFQ-25 and SF-36
Biological: Blood samples — Additional blood samples for immunomonitoring

SUMMARY:
Uveitis is characterized by inflammation of the uvea, which is the middle portion of the eye. The greatest challenge for the treatment of uveitis is patients who have inflammation involving the posterior segment, either primarily in the vitreous (intermediate uveitis), the choroid or retina (posterior uveitis), or involving the entire eye (panuveitis). The term "uveitis" denotes a heterogeneous collection of diseases including infections, systemic immune-mediated diseases like sarcoidosis, and immune-mediated syndromes confined to the eye like sympathetic ophthalmia. Despite the progress in recent decades, uveitis and the related intraocular inflammation are comparable to diabetes or macular degeneration as a cause of lost quality-adjusted life years due to visual morbidity, and as such are a significant public health problem. The Standardization of Uveitis Nomenclature Working Group Guidelines recommend the use of corticosteroids as the first-line therapy for patients with active uveitis. However, long-term corticosteroid treatment can cause serious systemic and ocular side effects, such as hypertension, diabetes, osteoporosis, cataract, and glaucoma that limit its use in the treatment of uveitis. Alternatively, immunomodulatory therapy (IMT) drugs are given as steroid-sparing agents and have shown good clinical results for both systemic diseases and ocular inflammatory diseases. Given the side effects of chronic corticosteroid therapy and better understanding of the mechanisms of autoimmune-mediated uveitis, the aim of the treatment for patients with noninfectious uveitis is steroid-free remission with IMT. While uveitis is a heterogeneous disease with polygenic and environmental factors, most forms of immune-mediated uveitis are thought to be due to an imbalance between regulatory mechanisms that inhibit the immune system and inflammatory mechanisms, which have evolved to rid the body of infectious organisms, but which can result in immune-mediated, often chronic disease if they are activated outside the context of the immediate infection. The pathophysiology of non-infectious uveitis involves the rupture of peripheral tolerance, resulting in auto-aggressive Th1 or Th17 lymphocytes reaching the eye. L-12 and IL-23 are two key cytokines involved in Th1 and Th17 polarization in uveitis, respectively. Furthermore, these two cytokines share a common subunit (p40). Ustekinumab, a humanized anti-p40 monoclonal antibody, is able to target both IL-12 and IL-23 pathways, thus disrupting Th1 and Th17 immune responses.

Decreasing the dose as well as the duration of treatment with GC is of particular importance in uveitis, and ustekinumab, which selectively inhibits Th1 and Th17 pathways in the inflammatory cascade, could provide a ideal additional therapy for non-infectious severe uveitis (NISU) to reach this objective.

Therefore, in the present study, we propose to evaluate the efficacy and safety of ustekinumab for the treatment of NISU.

ELIGIBILITY:
Inclusion criteria:

* Patients with newly diagnosed active NISU: evidence of activity within the 3 months prior to the screening visit as per:

  * VH (visual haze) ≥ 4 on the Miami 9-step scale (or VH >1+ according to SUN classification)
  * and/or macular edema on OCT (Central retinal thickness ≥ 300 microns)
  * and/or other signs of intraocular inflammation (e.g. perivascular sheathing of retinal vessels or leakage of retinal vessels on fluorescein angiography (FA)).
* Patients judged to be in good health as determined by the Principal Investigator based upon the results of medical history, laboratory profile, physical examination, chest x-ray (CXR), and a 12-lead electrocardiogram (ECG) performed during Screening.
* For men and women of childbearing age, effective contraception must be used by the patient and/or his/her partner throughout the duration of treatment with ustekinumab and until 23 weeks after the end of treatment. Breastfeeding is allowed 23 weeks after the end of treatment. Women considered without risk of pregnancy are those with :

  * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
  * progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
  * intrauterine device (IUD)
  * intrauterine hormone-releasing system ( IUS)
  * bilateral tubal occlusion
  * vasectomised partner
  * sexual abstinence
  * or those surgically sterile (bilateral oophorectomy or hysterectomy).
  * or at least one year of menopause (amenorrhea for at least 12 months)
* Patients over 18 years of age
* Affiliation to a the French health insurance system
* Patients who have given their consent

Exclusion criteria:

* Surgery scheduled within 12 months
* Patients with dementia
* Non-compliant patients
* Weight <45 kg or > 100 kg
* Patients under ward of court, tutelage or legal guardianship
* Pregnant or breast-feeding women

Exclusion criteria related to uveitis:

* Infectious uveitis, masquerade syndromes, or uveitis due to causes other than non-infectious uveitis disease (idiopathic uveitis is permitted)
* Isolated anterior uveitis
* Presence of cataract or posterior capsular opacification so severe that an assessment of the posterior segment of either eye is inadequate or impossible
* Contraindication to mydriasis in either eye or presence of posterior synechiae in the study eye such that mydriasis is inadequate for posterior segment examination
* Intraocular pressure ≥ 25mmHg by Goldmann tonometry or advanced glaucoma (e.g., cup-to-disc ratio > 0.9, split fixation on visual field, or need for > 3 intraocular pressure lowering medications to keep IOP < 22 mmHg) in either eye
* Monocular patient
* Sarcoidosis-related uveitis

Exclusion criteria related to ustekinumab:

* History of congenital or acquired immunodeficiency (e.g. common variable immunodeficiency disease).
* History of prior treatment with ustekinumab
* Hypersensitivity to ustekinumab, one of its excipients or another human or murine monoclonal antibody or latex
* Evidence of active infection at the time of baseline visit, or other Infectious contraindication to ustekinumab
* Neoplasia < 5 years, (except for in situ cervical cancer and skin carcinoma with R0 resection)
* Active tuberculosis or sign of latent tuberculosis (based on a history of untreated contact, a history of opacity of more than 1 cm in diameter on the chest x-ray, or an in vitro test positive[Quantiferon® or T-spot-TB®]). A history of TB disease or latent TB whose treatment was completed is not an exclusion criteria, regardless the Quantiferon® or T-spot-TB® is positive or not.
* Known positive laboratory test for syphilis serology, HIV antibody, hepatitis B surface antigen or anti-nucleocapsid antibody of hepatitis B virus, and/or hepatitis C antibody.
* History of multiple sclerosis and/or other demyelinating disorders
* Infection(s) requiring treatment with intravenous (IV) anti-infectives within 30 days prior to the Baseline Visit or oral anti-infectives within 14 days prior to the Baseline Visit.
* Screening laboratory and other analyses showing any of the following abnormal results:

  * AST, ALT > 1.75 × upper limit of the reference range;
  * WBC count < 3.0 × 109/L;

Other treatments:

* Corticosteroids

  * History of ≥3 systemic corticosteroid therapies (topical or inhaled treatments allowed) for another disease (e.g. asthma) within the last 6 months before screening visit
  * Dexamethasone intravitreal implant less than 6 months prior to study
* Patients receiving (or having stopped for less than 6 months or 5 elimination half-lives) an immunosuppressive or immunomodulatory drug or biotherapy:

  * anti TNF-α,
  * tocilizumab,
  * abatacept,
  * anakinra,
  * methotrexate,
  * azathioprine,
  * ciclosporine,
  * cyclophosphamide,
  * dapsone
  * or corticosteroid pulses
* Live vaccine administered within 30 days preceding inclusion
* Hypersensibility to fluorescein and indocyanin green

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Percentage of remission | Through study completion, an average of 30 months
Percentage of patients free of relapse between week 6 and week 24 | Through study completion, an average of 30 months

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CH Avignon, Avignon
  - CHU Dijon Bourgogne, Dijon